CLINICAL TRIAL: NCT04784650
Title: The Prevalence of Foot Complaints/Problems and Ulcers in a Pre-dialysis Population: a Cross-sectional Study
Brief Title: The Prevalence of Foot Complaints/Problems and Ulcers in a Pre-dialysis Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S64716
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Foot Ulcer; Diabetes Mellitus; Chronic Kidney Diseases; Pre-dialysis
MeSH Terms: conditions — Foot Ulcer; Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-dialysis population (Other): Pre-dialysis population, consisting both Diabetes Mellitus (DM) and non-DM patients
  Interventions: Other: Pre-dialysis population

INTERVENTIONS:
Other: Pre-dialysis population — Pre-dialysis population, consisting of both Diabetes Mellitus (DM) and non-DM patients

SUMMARY:
Diabetes mellitus is one of the main causes of chronic kidney disease (CKD) and an increased risk of foot complications is seen in patients suffering from both DM and CKD. CKD and DM patients share a trilogy of risk factors that contribute to the development of foot ulcers. This trilogy consists of peripheral arterial disease (PAD), neuropathy and an increased susceptibility to infection with an impaired wound healing. Additionally, almost one quarter of adults with CKD have to cope with depression.

The aim of our study is to determine the prevalence and types of foot problems in a pre-dialysis population, consisting of both DM and non-DM patients. If possible, risk factors will be determined. The detrimental effects of poor kidney function and foot problems on the quality of life and the general health status will be analyzed. A higher prevalence of PAD, peripheral neuropathy and DM are expected in patients with foot problems compared to those without.

DETAILED DESCRIPTION:
Plenty of research has been published regarding the prevalence of foot ulcers in a diabetes mellitus (DM) population. Zhang et al. concluded that foot ulceration is prevalent in 6,3% of DM patients worldwide. Moreover, diabetes mellitus is one of the main causes of chronic kidney disease (CKD) and an increased risk of foot complications is seen in patients suffering from both DM and CKD. Furthermore, dialysis treatment is also associated with a higher probability of foot ulceration.

According to Ndip et al., CKD and DM patients share a trilogy of risk factors that contribute to the development of foot ulcers. This trilogy consists of peripheral arterial disease (PAD), neuropathy and an increased susceptibility to infection with an impaired wound healing. Both diabetic and non-diabetic CKD patients have a high risk for peripheral neuropathy, creating a decreased sensation in the feet. This makes them more vulnerable for minor trauma, leading to the development of foot ulcers. These often precede more serious foot complications like infections and amputations, which have a great impact on the morbidity and mortality of the patient. They also cause a major financial load for the healthcare system.

Additionally, almost one quarter of adults with CKD have to cope with depression. This is independently associated with a reduced quality of life in a pre-dialysis population. The quality of life is also impaired by the presence of PAD, peripheral neuropathy and foot problems. Unfortunately, patients can be so overwhelmed by their renal disease that they avoid education and self-care, which can lead to even more complications and health costs.

In UZ Leuven, patients with a severe loss of kidney function (down to 25 percent or less of the normal function) are taken up in the pre-dialysis program. In contrast to DM and dialysis patients, there is a paucity of data about the prevalence of different foot problems in a pre-dialysis population. Freeman et al. performed one of the few studies that also include non-DM CKD patients. Hereby, a similar frequency of foot ulcers was found in CKD patients as in DM patients. However, an important limitation of the study is the small sample group size, so further research is needed. As CKD in stages 3 to 5 may affect approximately 10% of the global population, it is important to learn more about the different foot complaints that occur in these patients.

The aim of our study is to determine the prevalence and types of foot problems in a pre-dialysis population, consisting of both DM and non-DM patients. If possible, risk factors will be determined. The detrimental effects of poor kidney function and foot problems on the quality of life and the general health status will be analyzed. A higher prevalence of PAD, peripheral neuropathy and DM are expected in patients with foot problems compared to those without.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must counsel the pre-dialysis outpatient ward at UZ Leuven
* Minimum age of 18 years old
* Signed informed consent

Exclusion Criteria:

* Unable to understand Dutch
* Unable to fill in questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-04-24 (Actual)

PRIMARY OUTCOMES:
Presence of foot problems (no = 0, yes = 1) | at baseline
  To describe the prevalence and type of foot complaints/problems in a pre-dialysis population during foot assessment

SECONDARY OUTCOMES:
European Foot and Ankle Society (EFAS) questionnaire | at baseline
  To explore the possible risk factors that cause particular foot complaints/problems and to formulate suggestions to create a future prevention program to avoid, where possible, foot problems
Kidney Disease Quality of Life Short Form (KDQOL-SF) questionnaire | at baseline
  To evaluate the repercussion of these foot problems on the general health status and the quality of life of the patients
Indication of peripheral arterial disease (PAD) | at baseline
  Patient records will be screened for available medical imaging (in any form) of the blood vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Matricali, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No